CLINICAL TRIAL: NCT00870948
Title: Phase 1 BA Study, Single Center With Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Joaquin Valdes, MD, Abbott
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: M10-220
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Last update posted 2010-11-08 (Estimated); Status verified 2010-09

CONDITIONS: Healthy
Keywords: Open Label; Healthy Volunteers
MeSH Terms: interventions — briakinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Regimen A (Experimental): One 100 mg ABT-874 (pre-filled syringe liquid formulation from the 6000 L process) injected subcutaneously in the abdominal region at a 45 degree angle
  Interventions: Drug: ABT-874
- Regimen B (Experimental): One 100 mg ABT-874 (pre-filled syringe liquid formulation from the 6000 L process) injected IV in an arm vein
  Interventions: Drug: ABT-874
- Regimen C (Experimental): One 100 mg ABT 874 (reconstituted lyophilized powder from the 3000 L process) injected subcutaneously in the abdominal region at a 45 degree angle
  Interventions: Drug: ABT-874
- Regimen D (Experimental): One 100 mg ABT-874 (reconstituted lyophilized powder from the 1000 L process) injected subcutaneously in the abdominal region at a 45 degree angle
  Interventions: Drug: ABT-874
- Regimen E (Experimental): 700 mg ABT-874 (reconstituted lyophilized powder from the 3000 L process) in 100 mL 5% dextrose solution IV infusion in an arm vein
  Interventions: Drug: ABT-874

INTERVENTIONS:
Drug: ABT-874 — See Arm Description for details regarding specific Intervention Description that is attributed to each Arm, respectively.

SUMMARY:
Single dose in healthy volunteers to assess bioavailability (amount of study drug in the system) between different formulations of ABT-874.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be healthy

Exclusion Criteria:

* Subjects who are not healthy, enrolled in another study, or who have received ABT-874 previously.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2009-01; Primary Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Bioavailability following single dose | Hours: 0, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, 168, 240, 336, 504, 672, 1008, 1344 for Regimens A, C, D and additional hours 4 & 8 for Regimen B and hours 0.5 and 6 hours for Regimen E

SECONDARY OUTCOMES:
AEs, serious adverse events (SAEs), laboratory data, ADA and vital signs will be assessed throughout the study | Through Day 85 (and / or 45 days after study drug stoppped)

CONTACTS AND LOCATIONS:
Overall Officials: Joaquin Valdes, MD, Study Director — Abbott
Locations (1):
- Site Reference ID/Investigator # 16001, Evansville, Indiana, United States